

# TRIAL STATISTICAL ANALYSIS PLAN

c33744236-02

**BI Trial No.:** 1280-0022

Title: Xenera™ 1: A multi-centre, double-blind, placebo-controlled,

> randomised phase II trial to compare efficacy of xentuzumab in combination with everolimus and exemestane versus everolimus and exemestane in women with HR+ / HER2- metastatic breast

cancer and non-visceral disease

Including Protocol Amendment 5 < 1280-22 > -protocol-version-05

[c18323506-08]

**Investigational Product:** 

Xentuzumab (BI 836845)

Responsible trial statistician:



Phone:

**Date of statistical** analysis plan:

23 AUG 2021 SIGNED

2 Version:

**Page 1 of 37** 

Proprietary confidential information

© 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

8.

| Proprietar | y confidential information © 2021 Boenringer ingement international offion of one of more of its attributed | companies |
|---|---|---|
| 1. | TABLE OF CONTENTS | |
| TITLE | PAGE | 1 |
| 1. | TABLE OF CONTENTS | 2 |
| LISTO | F TABLES | |
| 2. | LIST OF ABBREVIATIONS | |
| 3. | INTRODUCTION | |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| <b>5.</b> | ENDPOINTS | |
| 5.1 | PRIMARY ENDPOINT | |
| 5.2 | SECONDARY ENDPOINTS | |
| <b>5.2.1 5.2.2</b> | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | 10 |
| 6. | GENERAL ANALYSIS DEFINITIONS | 19 |
| 6.1 | TREATMENTS | |
| <b>6.2</b> | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.3 | PATIENT SETS ANALYSED | 20 |
| 6.5 | POOLING OF CENTRES | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| | PLANNED ANALYSIS | |
| 7.<br>7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.1<br>7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4 | PRIMARY ENDPOINT | |
| 7.4.1 | Primary analysis of the primary endpoint | 26 |
| 7.5 | CECOND A DV ENDDOINTS | 25 |
| 7.5<br>7.5.1 | SECONDARY ENDPOINTS | |
| 7.5.1<br>7.5.2 | Secondary endpoints | |
| 7.5.2 | Secondary chaponics | |
| 7.7 | EXTENT OF EXPOSURE | 29 |
| <b>7.8</b> | SAFETY ANALYSIS | 30 |
| <b>7.8.1</b> | Adverse Events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs | |
| 7.8.4<br>7.8.5 | ElectrocardiogramOthers | |
| /.0.3 | Villers | 34 |

| <b>Boehringer Ingelheim</b> |
|-------------------------------|
| TSAP for BI Trial No: 1280.22 |

| c <b>3374</b> 4 | 12. | 36- | 02 |
|-----------------|-----|-----|----|
| Раде | 3 | Λf | 37 |

| 10. | HISTORY | TABLE | 3 |
|-----|----------|--------|---|
| 10. | IIISTOKI | 1 ADLE | , |

# LIST OF TABLES

| Table 5.1: 1 | Derivation rules for PFS | 9 |
|---|---|---|
| Table 5.2.2: 1 | Derivation rules for pain progression or intensification of pain palliation. | 11 |
| Table 6.2: 1 | Handling of iPDs | 20 |
| Table 6.7: 1 | Nominal time-points and windows for imaging | 24 |
| Table 6.7: 2 | Nominal time-points and windows for PROs | 24 |
| Table 7.8.1: 1 | Overview of Special Search Categories | 31 |
| Table 10: 1 | History table | 37 |

#### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|----------|-----------------------------------------------------------------|
| ADA | Anti-drug antibodies |
| AE | Adverse Event |
| ALT | Alanine aminotransferase |
| AQA | Analgesic Quantification Algorithm |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BI | Boehringer Ingelheim |
| BIcMQ | Boehringer Ingelheim customised MedDRA Queries |
| BOR | Best Overall Response |
| BPI-SF | Brief Pain Inventory – Short Form |
| CDK | Cyclin-Dependent Kinase |
| CI | Confidence Interval |
| COVID-19 | Coronavirus Disease 2019 |
| CR | Complete Response |
| CTC | Common Terminology Criteria |
| CTP | Clinical Trial Protocol |
| DC | Disease Control |
| DLM | Database Lock Meeting |
| DMC | Data Monitoring Committee |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| EQ-5D-5L | EuroQoL 5-dimension health status self-assessment questionnaire |
| HLT | High Level Term |
| HR | Hazard Ratio |
| ICH | International Conference on Harmonisation |
| iPD | Important Protocol Deviation |
| IRT | Interactive Response Technology |
| ITT | Intention-to-Treat |
| KM | Kaplan-Meier |
| Max | Maximum |

Min Minimum

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed Model Repeated Measures
MQRM Medical Quality Review Meeting

nAb Neutralising antibody

NFBSI-16 Network Functional Assessment of Cancer Therapy-Breast Cancer

Symptom Index

OR Objective response
OS Overall Survival

PD Progressive Disease

PFS Progression-free survival

PPS Per Protocol Set
PR Partial Response

PRO Patient Reported Outcome

PRO-CTCAE Patient Reported Outcomes-Common Terminology Criteria for Adverse

**Events** 

PT Preferred Term
Q1 Lower quartile
Q3 Upper quartile

RECIST Response Evaluation Criteria in Solid Tumours

RPM Report Planning Meeting

RS Randomised Set

SARS-CoV-2 Severe Acute Respiratory Syndrome Coronavirus 2

SD Stable Disease

SMQ Standardised MedDRA Query

SOC System Organ Class

SSC Special Search Categories

TFST Time to First Subsequent Therapy

TS Treated Set

TSAP Trial Statistical Analysis Plan

TSST Time to Second Subsequent Therapy

TTE Time to Event

ULN Upper Limit of Normal

WHO-DD World Health Organisation Drug Dictionary

### 3. INTRODUCTION

As per International Conference on Harmonisation (ICH) E9 guidance (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Trial Statistical Analysis Plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including protocol amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

This TSAP currently covers the Phase II part of the study, for the scenario that the criterion for expanding the trial seamlessly into Phase III has not been met. In such an instance, the trial will be unblinded and the results evaluated in an explorative manner to see if they are sufficient for further development of this compound in this indication.

SAS® Version 9.4 or a later version will be used for all analyses.

### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

The following changes to the statistical methods described in the CTP and subsequent amendments are detailed in this TSAP:

• Where considered appropriate, the potential impact of Coronavirus Disease 2019 (COVID-19) on the study will be assessed by producing additional summaries of disposition, protocol deviations, treatment compliance, efficacy, treatment exposure and adverse events (AEs). The start date for COVID-19 having an impact on the trial will be taken as the earliest date of a COVID-19 related protocol deviation, discontinuation due to COVID-19, onset of a severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) related AE or COVID-19 related global BI recruitment hold (17 MAR20).

## 5. ENDPOINTS

Time to event (TTE) endpoints, unless stated otherwise, will be calculated as follows:

For patients with 'event' as an outcome:

• TTE [days] = date of outcome – date of randomisation + 1

For patients with 'censored' as an outcome:

• TTE (censored) [days] = date of outcome – date of randomisation + 1

Derivations will be calculated in days but will be presented as months in the respective outputs [Months =  $(Days \times 12) / 365.25$ ].

All references to the Response Evaluation Criteria in Solid Tumours (RECIST) are according to Version 1.1 in combination with MD Anderson criteria (refer to Section 5.1 of the CTP for further details). Unless stated otherwise, all imaging-related endpoints detailed below will primarily be derived from blinded independent assessment data, derivations using investigator assessment data will also be performed but will be supportive in nature.

#### 5.1 PRIMARY ENDPOINT

The primary endpoint is progression-free survival (PFS) calculated as the time from randomisation until progressive disease (PD) according to RECIST or death from any cause, whichever occurs earlier. The date of PD will be based upon blinded independent assessment.

The rules to determine the PFS outcome (event or censored) along with the date of outcome are specified in <u>Table 5.1: 1</u>. These rules will be applied to the independent assessment data prior to analysis.

In order to identify whether radiological imaging assessments are missing, a nominal time-point based on the scheduling detailed in the CTP will be assigned to each assessment according to <u>Table 6.7: 1</u>. If a patient does not have an assessment for one of the scheduled time-points, it will count as a missed assessment. Any assessment with an overall tumour

response of Not Evaluable (NE) will be considered as a missed assessment and cannot be used as an outcome date.

Derivation rules for PFS Table 5.1: 1

| Status at time of analysis | Outcome | Date of outcome |
|---|---|---|
| No baseline radiological assessment and/or no post-baseline radiological assessments | | |
| Death on or before the second planned radiological assessment | Event* | Date of death |
| Vital status is unknown or alive or death after second radiological assessment | Censored | Date of randomisation |
| With baseline and at least one post-baseline r | adiological a | ssessment |
| Alive and non-PD, no more than one consecutively missed radiological assessment | Censored* | Date of last radiological assessment |
| Alive and non-PD, two or more consecutively missed radiological assessments | Censored* | Date of last radiological assessment prior to missed radiological assessments |
| PD, no more than one consecutively missed radiological assessment prior to PD | Event* | Date of radiological assessment of PD |
| PD, two or more consecutively missed radiological assessments prior to PD | Censored* | Date of last radiological assessment prior to missed radiological assessments |
| Death and non-PD, no more than one consecutively missed prior radiological assessment prior to death | Event* | Date of death |
| Death and non-PD, two or more consecutively missed radiological assessments prior to death | Censored* | Date of last radiological assessment prior to missed radiological assessments |
| Initiation of subsequent anti-cancer therapy | | |
| Subsequent anti-cancer therapy started before the outcomes flagged with a '*' above | Censored | Date of last radiological<br>assessment before<br>subsequent anti-cancer<br>therapy (or date of<br>randomisation if none exist) |

<sup>\*</sup>For these outcomes if initiation of subsequent anti-cancer therapy occurred prior to the outcome date then the rule for the final row of table will be used instead

#### 5.2 **SECONDARY ENDPOINTS**

#### 5.2.1 **Key secondary endpoints**

There are no key secondary endpoints defined for the trial.

# 5.2.2 Secondary endpoints

#### Overall survival

Overall survival (OS) will be calculated as the time from randomisation to death from any cause. Patients without evidence of death will be censored at the date of last contact when known to be alive.

# Disease control

Disease control (DC), defined as a best overall response (BOR) of complete response (CR), partial response (PR), stable disease (SD) or Non-CR/Non-PD. SD and Non-CR/Non-PD must have been observed up until at least the Week 24 tumour assessment.

BOR is defined according to RECIST based on all evaluable tumour assessments from randomisation until the earliest of PD, start of subsequent anti-cancer therapy, loss to follow-up, withdrawal of consent or death. To be aligned with the primary endpoint derivation, tumour assessments after two or more consecutively missed assessments will not be considered.

### Duration of disease control

Duration of DC will be calculated as the time from randomisation until the earliest of PD (according to RECIST) or death from any cause, among patients with DC.

The outcome rules defined in <u>Table 5.1: 1</u> will be used for the calculation.

### Objective response

Objective response (OR), defined as a BOR (as detailed for DC) of CR or PR.

# Time to pain progression or intensification of pain palliation

Time to pain progression or intensification of pain palliation, defined as the time from randomisation until the earliest of:

- ≥2 point increase from baseline in the Brief Pain Inventory Short Form (BPI-SF), Item 3 (worst pain), without a decrease (of ≥1 point) from baseline analgesics use (via the 8-point Analgesic Quantification Algorithm [AQA]), or
- $\geq$ 2 point increase from baseline in the AQA, or
- Death

The rules to determine outcome (event or censored) along with the date of outcome are specified in <u>Table 5.2.2: 1</u>. These rules will be applied to the independent assessment data prior to analysis.

In order to identify whether questionnaire assessments are missing, a nominal time-point based on the scheduling detailed in the CTP will be assigned to each assessment according to <u>Table 6.7: 2</u>. If a patient does not have an assessment for both the BPI-SF, Item 3 and the AQA score at one of the scheduled time-points, it will count as a missed assessment;

otherwise, a response will be derived. If a  $\geq 2$  point increase from baseline in the BPI-SF, Item 3 is observed but the AQA score is missing, it will be assumed that no decrease in analgesics use has taken place.

Table 5.2.2: 1 Derivation rules for pain progression or intensification of pain palliation

| Status at time of analysis | Outcome | Date of outcome |
|---|---|---|
| No baseline assessment and/or no post-baseline assessments | | |
| Death on or before the second planned assessment | Event* | Date of death |
| Vital status is unknown or alive or death after second planned assessment | Censored | Date of randomisation |
| With baseline and at least one post-baseline a | ssessment | |
| Alive and event-free, no more than one consecutively missed assessment | Censored* | Date of last assessment |
| Alive and event-free, two or more consecutively missed assessments | Censored* | Date of last assessment prior to missed assessments |
| Alive with event, no more than one consecutively missed assessment prior to event | Event* | Date of assessment of event |
| Alive with event, two or more consecutively missed assessments prior to event | Censored* | Date of last assessment prior to missed assessments |
| Death and event-free, no more than one consecutively missed assessment prior to death | Event* | Date of death |
| Death and event-free, two or more consecutively missed assessments prior to death | Censored* | Date of last assessment prior to missed assessments |
| Initiation of subsequent anti-cancer therapy | | |
| Subsequent anti-cancer therapy started before outcomes flagged with a '*' above | Censored | Date of last assessment<br>before subsequent anti-<br>cancer therapy (or date of<br>randomisation if none exist) |

<sup>\*</sup> For these outcomes if initiation of subsequent anti-cancer therapy occurred prior to the outcome date then the rule for the final row of table will be used instead









### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For reporting purposes, all randomised patients will be classified into either 'Xe1000+Ev10+Ex25' or 'Plc+Ev10+Ex25' as randomised. For efficacy analyses, the intent-to-treat (ITT) approach will be used, i.e. patients will be analysed according to the treatment group they were randomised to. All planned analyses will be presented by this randomised treatment group. Handling of patients where treatment group assignment has not been followed will be handled on a case-by-case basis, to be agreed at report planning meetings prior to database lock. The following study periods are defined:

- Screening: day of informed consent to day prior to first administration of study treatment
- Treatment: day of first administration of study treatment to day of last administration of study treatment
- Residual effect period (REP): day after last administration of study treatment, for a duration of 42 days
- Follow-up: day after the end of the REP to trial completion

For safety analyses, treated patients will be analysed according to the initial treatment taken, and for safety summaries, data recorded whilst taking study treatment and up to 42 days after last administration of study treatment (i.e. including the REP) will be considered as ontreatment. As the treatment arms are made up of a combination of individual treatments, a patient may have multiple last doses of treatment; therefore, the last dose of study medication is defined as the latest of these.

### 6.2 IMPORTANT PROTOCOL DEVIATIONS

No per protocol set (PPS) analysis will be performed, hence, no patient will be excluded from the analyses (with the exception of patients not providing informed consent). However, patients with potentially important protocol deviations (iPDs) will be documented to give an indication of the level of adherence to the protocol, refer to <a href="Table 6.2:1">Table 6.2:1</a>. Note this is a working list and may not be finalised until the final Medical Quality Review Meeting (MQRM), Database Lock Meeting (DBLM) and Report Planning Meeting (RPM) have taken place prior to the database lock of the primary PFS analysis.

A frequency table of the above iPDs will be produced. In addition, a frequency table of all COVID-19 related non-important and important PDs will be produced.

Table 6.2: 1 Handling of iPDs

| iPD code | iPD Category & Brief Description | Analysis Set Excluded from |
|---|---|---|
| A1 | Diagnosis of trial disease questionable | None |
| A2 | Prohibited baseline condition, diagnosis or treatment | None |
| A3 | Laboratory result indicating inadequate organ function at screening | None |
| A4 | Adequate archival tumour tissue not available | None |
| B1 | Informed consent not available/not done | All |
| B2 | Informed consent too late | None |
| В3 | Age limit for patient inclusion not adhered to | None |
| C1 | Time window violation for procedures performed at screening | None |
| C2 | Trial medication not given according to protocol | None |
| С3 | Infusion time for the investigational treatment outside of CTP specific boundaries | None |
| C4 | Randomisation not followed | None |
| D1 | Prohibited treatment during trial conduct phase | None |
| E1 | Imaging assessments not done according to CTP instructions | None |
| F1 | Other protocol violations affecting patient rights or safety | None |

### 6.3 PATIENT SETS ANALYSED

The following patient sets are defined:

### • Enrolled set:

This patient set includes all patients who have given informed consent. The enrolled set will be used for patient disposition summaries.

## • Randomised set (RS):

This patient set includes all randomised patients, regardless of whether they have received treatment or not. The RS will be used for demographic and baseline characteristic summaries and the evaluation of primary, secondary and further endpoints.

- Treated set (TS):
  - This patient set includes all patients who are documented to have received and taken at least one dose of any study medication. The TS will be used for the evaluation of safety.
- PK parameter analysis set (PKS): This patient set includes all patients in the TS who have at least one valid drug plasma concentration available that was not excluded because of protocol deviations affecting PK evaluation.





#### 6.5 POOLING OF CENTRES

This section is not applicable because centre is not included in the statistical model.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

In general, missing data will not be imputed, unless required for the following analyses and definitions. Then the rules as described below apply.

For TTE endpoints, patients who are event-free but have dropped out of the trial prematurely or are not evaluable for other reasons will be censored according to the rules given in <u>Sections</u> <u>5.1</u>, <u>5.2</u> and <u>5.3</u>.

The BPI-SF pain interference aggregated score will only be calculated if 4 or more of the 7 individual item scores have been completed.

Missing or incomplete dates that affect the evaluation of endpoints will be imputed utilising a worst-case approach, which will be applied on a case-by-case basis (depending on the affected endpoint) and documented appropriately prior to database lock and unblinding.

For the purposes of potential PFS censoring incomplete start dates of subsequent anti-cancer therapy will be imputed. The earliest possible date will be assumed, if this results in a start date prior to the stop date of study treatment this will be defaulted to study treatment stop date + 1 day.

Missing or incomplete adverse event (AE) dates will be imputed according to BI standards (2).

For the calculation of time to first diagnosis, if the date of diagnosis is incomplete the 1<sup>st</sup> will be used for a missing day and January for a missing month.

In general, actual patient data as reported in the eCRF will be used for analyses. If the data relating to the assignment of stratification factors are missing in the eCRF then the values entered into the Interactive Response Technology (IRT) system will be used instead (note these entries are automatically transferred to the eCRF).

# 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The last measurement observed prior to start of trial medication will be assigned to baseline. Note that for some trial procedures this may be the value measured on the same day trial medication was started. In these cases, where time of measurement is not recorded, it will be assumed that the measurements were taken prior to the intake of any study medication.

For measurements where not only the examination date but also time are recorded, examination time will be taken into account when defining baseline. Therefore, a measurement recorded on the same date as the first study drug administration will be considered as the baseline value, if and only if, the recording time was before or the same as the time of first study drug administration. If any of these times are missing and the date of the measurement is equal to the date of first study drug administration, then the measurement will be considered according to what was planned in the protocol, i.e. for safety laboratory data prior to first study medication. Note this rule will be relaxed for PRO data, as long as the baseline assessment of PROs is performed on or prior to the date of first study drug administration it will be considered as a valid baseline.

For tumour assessments, baseline evaluations must be performed no more than 28 days prior to start of trial medication.

Study days and visits will be labelled according to the flow chart of the CTP. In alignment with the CTP, study day will be calculated relative to the date of the first administration of study drug. The day prior to first administration of study drug will be 'Day -1' and the day of first administration of study drug will be 'Day 1'. Hence, 'Day 0' will not exist.

In order to identify whether consecutive imaging time points are missing for a patient a nominal time point [8, 16, 24 weeks and every 8 weeks thereafter up to 80 weeks, and every 12 weeks thereafter] will be assigned to each image. This will be achieved by creating time windows for each assessment as detailed in Table 6.7: 1 below. If a patient does not have an image in one of the time windows when one is expected they will be considered as having 'missed an assessment' for that time-point. In case a patient has more than one assessment in one window, the assessment with the latest outcome will be used for the analysis unless progressive disease (PD) has been recorded earlier then PD will be used. Additionally, if a patient has multiple imaging dates within an assessment (e.g. a different target lesion imaging date to the non-target lesion imaging date), if the overall response is PD the earliest imaging date will be used, otherwise the latest imaging date will be used. Note for the slotting of imaging data and the derivation of time to efficacy events in general, 'Day 1' will be considered as the day of randomisation.

Table 6.7: 1 Nominal time-points and windows for imaging

| Nominal time-point<br>[Weeks] | Nominal time-point [Days] | Window [Days] |
|---|---|---|
| 0 | 1 | <=1 |
| 8 | 57 | [2, 85] |
| 16 | 113 | [86, 141] |
| +8 weeks* | +56 days* | [+56 days, +56 days]* |
| 80 | 561 | [534, 603] |
| 92 | 645 | [604, 687] |
| +12 weeks* | + 84 days* | [+84 days, +84 days]* |

<sup>\*</sup> For subsequent visits, add value to previous record in respective column

In a similar fashion to imaging time points, missed PRO assessments will be identified as detailed in Table 6.7: 2.

Table 6.7: 2 Nominal time-points and windows for PROs

| Nominal time-point<br>[Weeks] | Nominal time-point [Days] | Window [Days] |
|---|---|---|
| 0 | 1 | <=1# |
| 4 | 29 | [2, 43] |
| 8 | 57 | [44, 71] |
| +4 weeks* | +28 days* | [+28 days, +28 days]* |
| 80 | 561 | [548, 589] |
| 88 | 617 | [590, 645] |
| +8 weeks* | +56 days* | [+56 days, +56 days]* |

<sup>\*</sup> For subsequent visits, add value to previous record in respective column

Note if a patient discontinues study treatment and enters the follow-up for progression then PRO assessments will follow the imaging assessment schedule, so will either be 8-weekly or 12-weekly dependent upon whether reached Week 80 (Cycle 20) or not.

<sup>#</sup> Note any Course 1, Visit 1 data recorded prior to starting study medication will be defaulted to Day 1 even if it was after the randomisation date

### 7. PLANNED ANALYSIS

In general (unless specified elsewhere), BI standards (3) will be followed for the End-Of-Text tables. In summary:

- The set of statistics for continuous data is N / Mean / Standard Deviation / minimum (Min) / lower quartile (Q1) / Median / upper quartile (Q3) / Maximum (Max). Other than the Min and Max, all statistics will be presented to one more decimal place than the raw data.
- Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category 'missing' will only be displayed if there are actually missing values.
- Time-to-event endpoints will be summarised in months [Months = (Days x 12) / 365.25] to one decimal place. Hazard ratios (HRs) and corresponding confidence intervals (CIs) will be presented to two decimal places. P-values will be presented to four decimal places.

### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, for the RS of patients.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report, for the RS of patients.

Concomitant diseases will be coded using the most current version of Medical Dictionary for Regulatory Activities (MedDRA) and will be summarised by primary system organ class (SOC) and preferred term (PT). Concomitant medications will be coded using the most current version of WHO-DD and will be summarised by ATC3 class and PT. In situations where a therapy belongs to more than one ATC3 class all classes will be presented, along with explanatory footnotes. Separate summaries of concomitant medications started prior to and during the period of taking study medication will be produced.

### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report, for the TS of patients. Appropriate summaries of compliance before and from the start of the COVID-19 disruption will also be produced.

### 7.4 PRIMARY ENDPOINT

The primary endpoint of PFS as assessed by blinded independent assessment will be analysed using the RS of patients.

# 7.4.1 Primary analysis of the primary endpoint

The primary endpoint will be analysed using a stratified (presence of baseline bone-only metastases, prior CDK4/6 inhibitor treatment, menopause status) log-rank test to assess the effect of treatment.

A stratified Cox proportional hazards model will be used to estimate the HR of the treatment effect and the corresponding asymptotic two-sided 95% Wald CI. A HR of less than one will favour the xentuzumab arm. Breslow's method for handling ties will be used.

Kaplan-Meier (KM) estimates will be used to display the distribution of PFS for each treatment group on a KM curve. To support the plot, estimated survival probabilities at specific time points of interest (scheduled imaging time-points) will be tabulated along with 95% CIs, using Greenwood's variance estimate. In addition, the survival distribution will be used to provide estimates of the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles.

Suitable methods will be used to check the assumption of proportional hazards.





#### 7.5 SECONDARY ENDPOINTS

# 7.5.1 Key secondary endpoints

This section is not applicable, as no key secondary endpoint has been specified in the protocol.

# 7.5.2 Secondary endpoints

# Overall survival

The analysis of this endpoint will follow that of the primary endpoint, detailed in <u>Section 7.4.1</u>.

# Disease control

A logistic regression model adjusting for the previously defined stratification factors will be used for the analysis of this binary endpoint. The treatment groups will be compared via the likelihood ratio test and presented along with the corresponding odds ratio and 95% CI. An odds ratio greater than one will favour the xentuzumab arm.

# Duration of disease control

KM estimates will be calculated for each treatment group to provide estimates of the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles and their corresponding 95% CIs.

# Objective response

OR will be analysed as for DC above.

# Time to pain progression or intensification of pain palliation

The analysis of this endpoint will follow that of the primary endpoint, detailed in Section 7.4.1.





#### 7.7 EXTENT OF EXPOSURE

A descriptive summary of total duration of study treatment will be produced both for the combined treatment and for each of the individual components. A dose reduction summary of everolimus will also be produced along with dose intensity summaries for each of the individual components of the study treatment. Refer to Section 5.4.2 for further details.

A Kaplan-Meier plot of the time to permanent discontinuation of all study medication (date of last administration of study medication – date of first administration of study medication + 1) will also be produced by treatment group. Patients who have not permanently discontinued study medication will be censored at the date of the snapshot for the analysis.

Appropriate summaries of exposure before and from the start of the COVID-19 disruption will also be produced.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set. In addition to the summaries described below, standard tables required for the clinical trials disclosure process (ClinicalTrials.gov and EudraCT) will be produced (4).

#### 7.8.1 Adverse Events

AEs will be coded with the most recent version of the MedDRA. The severity of AEs will be scaled according to Common Terminology Criteria (CTC) AE version 5.

Unless otherwise specified, the analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of patients with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the eCRF will be collapsed into an AE if all of the following applies:

- All AE attributes are identical (Lowest Level Term [LLT], CTCAE grade, action taken with trial medication, therapy required, seriousness, reason for seriousness, relationship, outcome, AE of special interest)
- The occurrences are time overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence).

For further details on the analysis and presentation of AE data refer to BI standards (5).

The analysis of AEs will be based on the concept of treatment emergent adverse events. That means that all AEs with an onset between first drug intake and last drug intake + REP (42 days) will be assigned to the randomised treatment. All AEs with an onset before first drug intake will be assigned to 'screening' and all AEs with an onset after the residual effect period will be assigned to 'post-treatment' (for listings only). For details on the treatment definition, see Section 6.1.

An overall summary of AEs will be presented; along with the standard categories presented additional categories for action taken and drug relationship with each compound, worst CTCAE grade and infusion related reaction response. The frequency of patients with AEs will be summarised by treatment, highest CTCAE grade, primary SOC and PT. The SOCs will be sorted alphabetically; PTs will be sorted by decreasing frequency (within SOC). Only AEs with a given CTCAE grade will be displayed in tables showing AEs by worst CTCAE grade. AEs with a missing CTCAE grade will not be displayed in these tables; a footnote will explain that these AEs are not included and a separate listing of them will be produced if required. The following tables will be produced for AEs during the on-treatment period:

- Patients with AEs
- Patients with any related AE

- Patients with related xentuzumab/placebo AEs
- Patients with related everolimus AEs
- Patients with related exemestane AEs
- Patients with SAEs
- Patients with related xentuzumab/placebo SAEs
- Patients with related everolimus SAEs
- Patients with related exemestane SAEs
- Patients with other significant AEs, defined as serious and non-serious AEs that lead to dose reduction or permanent discontinuation of any study medication
- Patients with AEs leading to death (no CTCAE grade required)
- Patients with AEs leading to discontinuation of xentuzumab/placebo
- Patients with AEs leading to discontinuation of everolimus
- Patients with AEs leading to discontinuation of exemestane
- Patients with AEs leading to dose reduction of everolimus
- Patients with AEs leading to dose interruption of xentuzumab/placebo
- Patients with AEs of Special Interest (refer to Section 5.2.6.1 of the CTP)

In addition some AEs are considered to be of particular importance and special search categories (SSC) of groupings of PTs based on Standardised MedDRA Queries (SMQ), BI customised MedDRA Queries (BIcMQ) or MedDRA High Level Terms (HLT) are defined at the project level, the latest version of which will be used. Details of the current version are provided in the Table 7.8.1: 1 below.

SSCs summaries of patients with AEs and related AEs by treatment, highest CTCAE grade, grouped term and PT will be produced. Similar summaries will be produced for the BIcMQ SARS-COV-2-infections.

Table 7.8.1: 1 Overview of Special Search Categories

| Grouped term | Groupings |
|---|---|
| Hepatic impairment | SMQ: Drug related hepatic disorders – comprehensive search |
| Hyperglycaemia narrow | SMQ: Hyperglycaemia / new onset diabetes mellitus (narrow terms only) |
| Infusion related reaction | SMQ: Hypersensitivity |
| Non-infectious pneumonitis | SMQ: Interstitial lung disease (narrow terms only) |
| Renal insufficiency | SMQ: Acute renal failure, SMQ: Proteinuria, HLT: Glomerulonephritis and nephrotic syndrome |
| Weight loss | BIcMQ: Weight loss |
| Neutropenia | SMQ: Haematopoietic leukopenia (narrow terms only) |
| Stomatitis | BIcMQ: Gastrointestinal mucositis (subsearch1: Stomatitis) |

Table 7.8.1: 1 Overview of Special Search Categories (cont.)

| Grouped term | Groupings |
|---|---|
| Asthenia | MedDRA PTs of Asthenia, Fatigue, Lethargy, Malaise, and Decreased activity |
| Haemorrhage | SMQ: Haemorrhage laboratory terms (narrow terms only), SMQ: Haemorrhage terms (excl. laboratory terms) |
| Anemia | SMQ: Haematopoietic erythropenia |
| Thrombocytopenia | SMQ: Haematopoietic thrombocytopenia (narrow terms only) |
| Thromboembolism | SMQ: Embolic and thrombotic, vessel type unspecified and mixed arterial and venous |
| Bradycardia | SMQ: Torsade de pointes/QT prolongation, PT of Bradycardia |
| Rash | BIcMQ: Skin eruptions (subsearch2: Skin rash potentially related to drug use) |

# 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (6). The same on-treatment periods as considered for the analysis of AEs will be applied for laboratory values. Patients having at least one post-baseline laboratory value will be displayed in the descriptive analyses.

The focus of the laboratory data analysis will be on the following primary laboratory parameters:

 Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, glucose, creatinine, platelets, cholesterol, triglycerides, neutrophils, lymphocytes, haemoglobin and white blood cells.

Descriptive statistics including baseline, last value on-treatment and change from baseline to last value on-treatment will be produced. CTCAE grades for applicable laboratory parameters will be calculated according to CTCAE version 5. The following outputs will be presented for each of the above parameters:

- Transitions of CTCAE grade from baseline to worst on-treatment laboratory value
- Transitions of CTCAE grade from baseline to last on-treatment laboratory value

Patients with no CTCAE grade due to missing laboratory values will be displayed as 'Missing'. Note with version 5 of the CTCAE grading some of laboratory parameters detailed above (ALT, AST and total bilirubin) can no longer be assigned a grade at baseline. For these parameters, the CTCAE shift tables will be replaced by shift tables of pre-defined categories

based on Upper Limit of Normal (ULN) values. A similar approach will also be adopted for creatinine due the ambiguity of CTCAE grading for grades 2 and 3. The pre-defined categories will follow BI standards (7).

Possible clinically significant abnormal laboratory values are defined as those laboratory values that are of CTCAE Grade  $\geq 2$  and show an increase from baseline value by at least one CTCAE grade. For those parameters for which no CTCAE has been defined, BI standard definition will be used to determine possible clinical significance. Frequency of patients with possible clinically significant abnormal laboratory values will be provided whenever applicable. If no baseline value is available (or CTCAE grading at baseline cannot be assigned) but the patient has a post-baseline laboratory value of CTCAE Grade  $\geq 2$  an increase from baseline will be assumed, i.e. the laboratory value considered as possible clinically significant.

#### Hepatic enzyme elevations (potential Hy's law cases):

The assessment of hepatic enzyme elevations will include frequencies of patients falling into the following categories:

- ALT and/or AST  $\geq$  3 x ULN with total bilirubin  $\geq$  1.5 x ULN
- ALT and/or AST  $\geq 3$  x ULN with total bilirubin  $\geq 2$  x ULN
- ALT and/or AST  $\geq$  3 x ULN with total bilirubin  $\geq$  2 x ULN and alkaline phosphatase  $\geq$  2 x ULN
- ALT and/or AST  $\geq$  3 x ULN with total bilirubin  $\geq$  2 x ULN and alkaline phosphatase < 2 x ULN
- Maximum ALT:  $\geq 3$ ,  $\geq 5$ ,  $\geq 10$  and  $\geq 20$  x ULN
- Maximum AST:  $\geq 3, \geq 5, \geq 10$  and  $\geq 20$  x ULN
- Maximum ALT and AST:  $\geq 3$ ,  $\geq 5$ ,  $\geq 10$  and  $\geq 20$  x ULN
- Maximum total bilirubin:  $\geq 1.5$  and  $\geq 2$  x ULN
- Maximum alkaline phosphatase:  $\geq 1.5$  and  $\geq 2$  x ULN

Where applicable for defining the above, events can occur in any order, but must occur within 30 days of each other, with an increase of either ALT or AST being the trigger for evaluations. Along with summaries of the above supportive eDISH plots will also be produced.

# 7.8.3 Vital signs

Only descriptive statistics are planned for this section of the report.

In order to investigate potential bradycardia a shift table of heart rate (<60 bpm,  $\ge60$  bpm) at baseline by lowest and last on-treatment heart rate (<60 bpm,  $\ge60$  bpm) will be produced. Other suitable summaries may be produced to investigate potential bradycardia.

# 7.8.4 Electrocardiogram

Electrocardiogram (ECG) results will only be listed; any clinically significant abnormalities will be recorded as either a concomitant diagnosis or an AE.

# **7.8.5** Others

Not applicable.

#### 8. **REFERENCES**

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|---|
| 2. | BI-KMED-BDS-HTG-0035: "How to Guide: Handling of Missing and Incomplete AE dates" |
| 3. | BI-KMED-BDS-HTG-0045: "How to Guide: Standards for Reporting of Clinical Trials and Project Summaries" |
| 4. | BI-KMED-BDS-QRG-0010: "Quick Reference Guide: Preparation of tables for results disclosure |
| 5. | BI-KMED-BDS-HTG-0066: "How to Guide: Analysis and Presentation of Adverse Event Data from Clinical Trials" |
| 6. | BI-KMED-BDS-HTG-0042: "How to Guide: Handling, Display and Analysis of Laboratory Data" |
| 7. | BI-KMED-BDS-HTG-0036: "How to Guide: CTCAE Grading for Laboratory Values" |

# 10. HISTORY TABLE

Table 10: 1 History table

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| 1 | 06-OCT-20 | | None | This is the final TSAP |
| 2 | 23-AUG-21 | | 5.2.2 | Clarified the minimum duration of DC. |
| | | | 6.7 | Allowing baseline PRO assessments measured on the same day of starting study treatment. |
| | | | 7.8.1 | Additional AE table added for 'any related' AEs. Update to SSCs. |



### APPROVAL / SIGNATURE PAGE

Document Number: c33744236 Technical Version Number: 2.0

**Document Name:** 8-01-tsap

**Title:** XeneraTM 1: A multi-centre, double-blind, placebo-controlled, randomised phase II trial to compare efficacy of xentuzumab in combination with everolimus and exemestane versus everolimus and exemestane in women with HR+/HER2-metastatic breast cancer and non-visceral disease

# **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|-------------------------------|-----------|------------------------|
| Approval-Project Statistician | | 23 Aug 2021 11:45 CEST |
| Approval | | 23 Aug 2021 17:23 CEST |
| Approval | | 23 Aug 2021 23:01 CEST |
| Approval | | 24 Aug 2021 16:48 CEST |
| Author-Trial Statistician | | 24 Aug 2021 16:52 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c33744236Technical Version Number: 2.0

# (Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|